CLINICAL TRIAL: NCT06869967
Title: Evaluation of Ultrasound-Guided Auricularis Magnus Nerve Block for Postoperative Pain Control in Ear Surgery
Brief Title: Evaluation of Postoperative Pain Control in Ear Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Nur Nazire Yucal, Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-KAEK-11
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain; Analgesia
Keywords: Regional Anesthesia; Ear Surgery; Auricularis Magnus Nerve Block
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricularis Magnus Nerve Block (Active Comparator): Ultrasound (US) -guided Auricularis Magnus Nerve Block with 5 ml 0.5 % bupivacaine will performe preoperatively to all patients in the AMG group.
  Interventions: Procedure: Auricularis Magnus Nerve Block
- Control (Active Comparator): In the control group, patients will be administered intravenous analgesics of 1 gram paracetamol, 20 mg tenoxicam, and 8 mg ondansetron 30 minutes before the end of the operation, as stated in the patient protocol, during their follow-up after general anesthesia.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Auricularis Magnus Nerve Block — Auricularis Magnus Nerve block will be performed using 5 mL of %0.5 bupivacaine
  Arms: Auricularis Magnus Nerve Block
Procedure: Control Group — Intravenous analgesics 1 gram paracetamol, 20 mg tenoxicam, 8 mg ondansetron will be administered.
  Arms: Control

SUMMARY:
Middle ear surgery is the most popular procedure in ear, nose and throat surgery. Increased sympathetic stimulation after surgery can activate the sympathetic system, causing hypertension and increased heart rate. As a result of these clinical conditions, hemorrhage can occur, which can impair the quality of the surgical field, which is undesirable in middle ear surgery.Clinical studies should be conducted with auricularis magnus nerve block applied in the perioperative period in middle ear surgery and postoperative pain scores.

DETAILED DESCRIPTION:
Middle ear surgery is the most popular procedure in ear, nose and throat surgery. Increased sympathetic stimulation after surgery can activate the sympathetic system, causing hypertension and increased heart rate. As a result of these clinical conditions, hemorrhage can occur, which can impair the quality of the surgical field, which is undesirable in middle ear surgery.Ultrasound-guided auricularis magnus nerve block can be used as a potential solution to these problems. Ultrasound-guided peripheral nerve block can be visualized. It is appropriate and applicable to block a single distal nerve with a small dose of local anesthetic under ultrasound guidance. Ultrasound-guided blocking of the blocked area has reduced side effects with increased accuracy and accurate analgesic effect.

In middle ear microsurgery, the nerve innervation of the postauricular incision area may not primarily originate from the auricularis magnus. Therefore, clinical studies should be conducted with auricularis magnus nerve block applied in the perioperative period in middle ear surgery and postoperative pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CWD and Mastodectom
* Patients undergoing elective surgery
* ASA (American Society of Anesthesiologists) physical status classification I-II
* Patients over 18 years of age

Exclusion Criteria:

* Anticoagulant use
* Allergy to the drugs to be used
* ASA (American Society of Anesthesiologists) physical status classification IV-V
* Presence of infection in the area where the block will be applied
* Patient's refusal to accept the block application or inability to cooperate with the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | During the operation
  Intraoperative opioid consumption

SECONDARY OUTCOMES:
Morphine consumption | 1 hours after surgery(T1), 6 hours after surgery (T2), 12 hours after surgery (T3), 24 hours after surgery (T4)
  Postoperative morphine consumption
NRS Scores | 1 hours after surgery(T1), 6 hours after surgery (T2), 12 hours after surgery (T3), 24 hours after surgery (T4)
  NRS scores of the patients after the surgery (0=no pain, 10=worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)